CLINICAL TRIAL: NCT04508803
Title: Combination of HX008 And Niraparib in GErm-line-mutAted Metastatic Breast Cancer: a muLti-centEr Phase II Study
Brief Title: Combination of HX008 And Niraparib in GErm-line-mutAted Metastatic Breast Cancer
Acronym: CHANGEABLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Professor, Fudan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHANGEABLE
Record Dates: First submitted 2020-08-09; First posted 2020-08-11 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2020-06

CONDITIONS: Treatment Efficacy
Keywords: Anti-PD-1 Monoclonal Antibodies; PARP Inhibitors; Breast Cancer; Homologous Recombination Deficiency
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- The main research (Experimental): Patients diagnosed with HER2 negative metastatic breast cancer with BRCA1/2, PALB2, CHEK2 pathogenic/suspected pathogenic germline mutation are recruited.
  Interventions: Drug: HX008，Niraparib
- Ancillary Exploration research 1 (Experimental): Patients diagnosed with HER2 negative metastatic breast cancer with DDR gene (include ATM、ATR、BAP1、BARD1、BLM、BRIP1、CHEK1、CDK12、FANCA、FANCC、FANCD2、FANCE、FANCF、FANCM、MRE11A、NBN、PTEN、RAD50、RAD51C、RAD51D、WRN)pathogenic/suspected pathogenic germline mutation except BRCA1/2, PALB2 and CHEK2 are recruited.
  Interventions: Drug: HX008，Niraparib
- Ancillary Exploration research 2 (Experimental): Patients diagnosed with HER2 positive metastatic breast cancer with DDR gene pathogenic/suspected pathogenic germline mutation are recruited.
  Interventions: Drug: HX008，Niraparib，Trastuzumab
- Ancillary Exploration research 3 (Experimental): Patients diagnosed with brain metastases breast cancer with DDR gene pathogenic/suspected pathogenic germline mutation who has not undergone or progressed after brain radiotherapyare recruited.
  Interventions: Drug: HX008，Niraparib，Pyrrolitinib

INTERVENTIONS:
Drug: HX008，Niraparib — Subjects received intravenous HX008 at a fixed dose of 200mg, administered every 3 weeks, and 200mg of Niraparib orally per day.Every 3 weeks is a cycle.
  Arms: The main research
Drug: HX008，Niraparib — Subjects received intravenous HX008 at a fixed dose of 200mg, administered every 3 weeks, and 200mg of Niraparib orally per day.Every 3 weeks is a cycle.
  Arms: Ancillary Exploration research 1
Drug: HX008，Niraparib，Trastuzumab — Subjects received intravenous HX008 at a fixed dose of 200mg once every 3 weeks; 200mg Niraparib orally per day;Trastuzumab 8mg/kg in the first cycle and 6mg/kg after the first cycle intravenously once every 3 weeks; Every 3 weeks is a cycle.
  Arms: Ancillary Exploration research 2
Drug: HX008，Niraparib，Pyrrolitinib — HER-2 negative subjects received intravenous HX008 at a fixed dose of 200mg, administered every 3 weeks, and 200mg of Neirapali orally per day. Every 3 weeks is a cycle.
  Her-2 positive subjects received intravenous HX008 at a fixed dose of 200mg once every 3 weeks; 200mg Niraparib orally per day; Pyrrolitinib is taken orally at 400mg per day; Every 3 weeks is a cycle.
  Arms: Ancillary Exploration research 3

SUMMARY:
A number of anti-PD-1/L1 monoclonal antibodies have been approved for the treatment of various advanced tumors in the world, and many studies on anti-PD-1 /L1 monoclonal antibodies for breast cancer are also being carried out. HX008 (Taizhou Hanzhong Biomedical Co., Ltd.China) combined gemcitabine and cisplatin (GP) regimen for first-line treatment of advanced triple negative breast cancer has been shown good efficacy. On the other hand,HRD as the target of PARP inhibitor therapy in the treatment of breast cancer has a broad prospect, In HRD tumor patients, the use of PARPi can make obstacles of DNA damage repair(DDR), accumulation of DNA damage, thus promote the apoptosis of tumor cells. Several PARPi have been approved worldwide (including Olaparib, Rucaparib, Niraparib, Talazoparib, Veliparib) for the treatment of ovarian and/or breast cancer. Theoretically, PARPi and anti-PD-1 monoclonal antibody can play a synergistic mechanism. In this study, HX008 combined with Niraparib is designed to treat metastatic breast cancer patients with DDR gene (BRCA1/2, PALB2, CHEK2, ATM, ATR, BAP1, BARD1, BLM, BRIP1, CHEK1, CDK12, FANCA, FANCC, FANCD2, FANCE, FANCF, FANCM, MRE11A, NBN, PTEN, RAD50, RAD51C, RAD51D, WRN) pathogenic/suspected pathogenic germline mutation, so as to explore the possibility of more combined therapy for breast cancer to achieve better therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

1. Performance Status 0-1.
2. Life expectancy longer than 3 months.
3. Histological proven unresectable recurrent or advanced breast cancer.
4. For ehe main research: Patients with histopathologically diagnosed advanced (recurrent or metastatic) HER2-negative breast cancer with definite pathogenic/suspected pathogenic germline mutations in BRCA1/2, or PALB2, or CHEK2.
5. For ancillary exploration research 1: Patients with histopathologically diagnosed advanced (recurrent or metastatic) HER2-negative breast cancer with definite pathogenic/suspected pathogenic germline mutations in ATM, or ATR, or BAP1, or BARD1, or BLM, or BRIP1, or CHEK1, or CDK12, or FANCA, or FANCC, or FANCD2, or FANCE, or FANCF, or FANCM, or MRE11A, or NBN, or PTEN, or RAD50, or RAD51C, or RAD51D, or WRN.
6. For ancillary exploration research 2: Patients with histopathologically diagnosed advanced (recurrent or metastatic) HER2-positive breast cancer with definite pathogenic/suspected pathogenic germline mutations in BRCA1/2, or PALB2, or CHEK2, or ATM, or ATR, or BAP1, or BARD1, or BLM, or BRIP1, or CHEK1, or CDK12, or FANCA, or FANCC, or FANCD2, or FANCE, or FANCF, or FANCM, or MRE11A, or NBN, or PTEN, or RAD50, or RAD51C, or RAD51D, or WRN.
7. For ancillary exploration research 3: Patients with histopathologically diagnosed advanced (recurrent or metastatic) breast cancer with brain and with metastases definite pathogenic/suspected pathogenic germline mutations in BRCA1/2, or PALB2, or CHEK2, or ATM, or ATR, or BAP1, or BARD1, or BLM, or BRIP1, or CHEK1, or CDK12, or FANCA, or FANCC, or FANCD2, or FANCE, or FANCF, or FANCM, or MRE11A, or NBN, or PTEN, or RAD50, or RAD51C, or RAD51D, or WRN.
8. Not more than 2 - line chemotherapy regimens were received in the stage of recurrence and metastasis.Platinum-based or PARP1 inhibitor treatment may be accepted, but the patient must have no disease progression during or within 8 weeks of the end of platinum-based or PARP1 inhibitor treatment at the stage of recurrence and metastasis, and relapse within 12 months after the end of neoadjuvant/adjuvant therapy.
9. Patients with hormone-receptor-positive, HER2 negative must received at least first-line endocrine therapy and progress to the stage of recurrence or metastasis, or have disease recurrence or metastasis during adjuvant endocrine therapy or within 1 year after the end of adjuvant therapy.
10. At least one extracranial measurable disease according to the response evaluation criteria in solid tumor (RECIST 1.1).
11. All patients enrolled are required to have adequate hematologic, hepatic, and renal function
12. Women of childbearing age must have a pregnancy test (serum or urine) that is negative within 7 days of enrollment, and be willing to use an appropriate method of contraception during the study and 8 weeks after the last dose of the study drug.
13. Be able to understand the study procedures and sign informed consent.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Treatment with an investigational product within 4 weeks before the first treatment.
3. Subjects have any active autoimmune disease, history of autoimmune disease, or history of disease or syndrome requiring systemic steroid or immunosuppressive medication.
4. Subjects had a history of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency disorders.
5. Received chemotherapy, radiotherapy, targeted therapy and major surgery within 3 weeks before the first administration;Received endocrine therapy within 2 weeks prior to first administration.
6. Uncontrolled serious infection.
7. Patients with hypertension and uncontrolled hypertension with hypotensive drugs therapy (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg). Patients with grade I or above myocardial ischemia or myocardial infarction or arrhythmia (including QT interval ≥ 440 ms) or cardiac insufficiency.
8. Inability to swallow, gastrointestinal resection, chronic diarrhea and obstruction of the intestine, various factors which affect drug use and absorption.
9. Patients with active viral hepatitis B or C.
10. Patients with chronic obstructive pulmonary disease (COPD), or pulmonary fibrosis.
11. Have received prior treatment with anti-PD-1/PD-L1 drugs and PARP inhibitors;
12. Patient who has a history of psychotropic substance abuse and is unable to stop or have a history of mental disorders.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 12 weeks
  ORR is the percentage of participants with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1. CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 30 months
  Time from date of randomization to the date of death from any cause
Progression-Free Survival (PFS) | Up to approximately 30 months
  PFS defined as the time from the date of randomization to the first evidence of disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant does not have a complete baseline disease assessment, then the PFS time was censored at the date of randomization, regardless of whether or not objectively determined disease progression or death has been observed for the participant. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Clinical Benefit Rate (CBR) | Up to approximately 12 weeks
  Percentage of participants with complete response (CR) or partial response (PR) or stable disease (SD) lasting 24 weeks or longer as defined in RECIST 1.1.CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD = Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease: PD = At least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20% the sum must also demonstrate an absolute increase of at least 5 mm.
Duration of Response (DOR) | Up to approximately 10 months
  Time from the first documented response (CR or PR) to the first documented progression or death due to underlying cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer center, Shanghai, China